CLINICAL TRIAL: NCT07373704
Title: Optimal Cut-off Points of Respiratory Muscle Strength and Endurance to Discriminate Disability Status in Multiple Sclerosis
Brief Title: Respiratory Muscle Strength and Endurance Cut-Offs in Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet Kaan ALTUNOK, Lecturer, Selcuk University
Other Study IDs: SelcukU_PT_MS_RESP_ENDURANCE_1
Record Dates: First submitted 2026-01-15; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Respiratory Muscle Strength; Respiratory Muscle Endurance; Pulmonary Function; Maximal Inspiratory Pressure; Maximal Expiratory Pressure; Cut-Off Values; EDSS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Multiple Sclerosis: Individuals diagnosed with multiple sclerosis undergoing assessment of respiratory muscle strength, respiratory muscle endurance, pulmonary function, walking performance, fatigue, and quality of life to determine optimal cut-off values for discriminating disability status.
  Interventions: Other: Respiratory Muscle Strength and Endurance Assessment

INTERVENTIONS:
Other: Respiratory Muscle Strength and Endurance Assessment — Participants will undergo a comprehensive assessment of respiratory muscle function, including respiratory muscle strength measured by maximal inspiratory and expiratory pressures and respiratory muscle endurance evaluated using an incremental threshold loading protocol. Pulmonary function will be assessed by spirometry. These assessments will be conducted to determine optimal cut-off values of respiratory muscle strength and endurance for discriminating disability status in individuals with multiple sclerosis and to examine their associations with clinical outcomes.

SUMMARY:
Multiple sclerosis (MS) is a chronic and progressive autoimmune disease of the central nervous system characterized by inflammation, demyelination, and axonal degeneration. Depending on lesion localization and disease severity, individuals with MS may develop a wide range of neurological manifestations affecting motor and sensory functions.

Current evidence indicates that pulmonary function impairments may occur in individuals with MS even in the absence of overt respiratory symptoms. Compared with healthy individuals, people with MS have been reported to exhibit significantly reduced values in several respiratory parameters, particularly respiratory muscle strength. Moreover, these reductions appear to become more pronounced in parallel with increasing Expanded Disability Status Scale (EDSS) scores, regardless of disease duration. Indeed, previous studies have demonstrated that even individuals with MS who have mild disability levels (EDSS 0-4.5) experience significant declines in respiratory muscle strength, pulmonary function, and functional exercise capacity compared with healthy controls.

These findings suggest that the respiratory system may be affected not only in the advanced stages of MS but also during the early phases of the disease, with functional impairments emerging before clinically evident respiratory complaints arise. Despite this, the existing literature lacks studies that define clear, clinically applicable cut-off values for respiratory muscle strength and endurance that can discriminate disability levels in individuals with MS. This gap highlights the absence of objective criteria that clinicians can rely on for early detection and for planning targeted rehabilitation interventions.

The present study aims to address this gap by identifying optimal cut-off points for respiratory muscle strength and endurance in individuals with MS to facilitate early and accurate discrimination of disability status. By doing so, this research seeks to make an original contribution to the literature. The findings are expected to support the standardization of respiratory assessment processes in clinical practice, thereby improving patient quality of life and enhancing the efficiency of healthcare services. Furthermore, the results will provide a strong scientific basis for integrating respiratory function assessments into MS follow-up protocols and will offer a methodological framework for future intervention-oriented studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with multiple sclerosis,
* Aged 18 years or older,
* Able to communicate effectively (able to speak, understand, read, and comprehend Turkish),
* No relapse within the past three months,
* Clinically stable for at least the past one month,
* No participation in respiratory-based rehabilitation programs within the past six months,
* Voluntary participation in the study.

Exclusion Criteria:

* Presence of neurological disorders other than multiple sclerosis,
* Presence of autoimmune diseases other than multiple sclerosis (e.g., rheumatoid arthritis, type 1 diabetes mellitus, systemic lupus erythematosus),
* Presence of chronic cardiac or pulmonary diseases that may affect respiratory muscle strength or pulmonary function, such as chronic obstructive pulmonary disease (COPD), asthma, interstitial lung disease, or heart failure,
* Pregnancy or breastfeeding,
* Inability to comply with the testing procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years and older diagnosed with multiple sclerosis who are clinically stable, able to communicate effectively, and eligible for respiratory muscle strength and endurance assessments.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory Muscle Strength (Maximal Inspiratory and Expiratory Pressures) | Baseline
  Respiratory muscle strength will be assessed by measuring maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) using an electronic mouth pressure device. Optimal cut-off values of respiratory muscle strength for discriminating disability status will be determined based on EDSS levels.
Respiratory Muscle Endurance | Baseline
  Respiratory muscle endurance will be evaluated using an incremental threshold loading protocol. The highest load sustained for at least one minute and the endurance index will be used to determine optimal cut-off values for distinguishing disability status in individuals with multiple sclerosis.

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | Baseline
  Disability status will be assessed using the Expanded Disability Status Scale (EDSS), a widely used measure of neurological disability in multiple sclerosis. The EDSS score ranges from 0 to 10, with higher scores indicating greater disability. A score of 0 represents normal neurological function, while a score of 10 indicates death due to multiple sclerosis. EDSS will be used as the reference standard for discrimination analyses.
Pulmonary Function: Forced Expiratory Volume in 1 Second (FEV₁) | Baseline
  Forced Expiratory Volume in one second (FEV₁) will be assessed using spirometry and reported in liters and as a percentage of predicted values. FEV₁ reflects expiratory airflow and pulmonary function.
Pulmonary Function: Forced Vital Capacity (FVC) | Baseline
  Forced Vital Capacity (FVC) will be measured using spirometry according to standardized American Thoracic Society and European Respiratory Society guidelines. FVC represents the maximum volume of air that can be forcibly exhaled after full inspiration and will be reported in liters and as a percentage of predicted values.
Pulmonary Function: FEV₁/FVC Ratio | Baseline
  The ratio of Forced Expiratory Volume in one second to Forced Vital Capacity (FEV₁/FVC) will be calculated from spirometric measurements and used to assess ventilatory patterns.
Pulmonary Function: Peak Expiratory Flow (PEF) | Baseline
  Peak Expiratory Flow (PEF) will be measured using spirometry and reported in liters per second to assess maximal expiratory flow capacity.
Pulmonary Function: Forced Expiratory Flow at 25-75% of FVC (FEF₂₅-₇₅) | Baseline
  Forced Expiratory Flow between 25% and 75% of FVC (FEF₂₅-₇₅) will be assessed using spirometry as an indicator of mid-expiratory airflow and small airway function.
Walking Speed (Timed 25-Foot Walk Test) | Baseline
  Walking speed will be evaluated using the Timed 25-Foot Walk test and examined in relation to respiratory muscle strength and endurance measures.
Perceived Walking Ability (Multiple Sclerosis Walking Scale-12) | Baseline
  Perceived walking ability will be assessed using the Multiple Sclerosis Walking Scale-12 (MSWS-12), a 12-item patient-reported outcome measure of walking impairment in individuals with multiple sclerosis. The total score is transformed to a 0-100 scale, with higher scores indicating greater walking impairment and worse perceived walking ability. MSWS-12 scores will be analyzed as clinical correlates of respiratory muscle strength and endurance.
Fatigue (Modified Fatigue Impact Scale) | Baseline
  Fatigue will be assessed using the Modified Fatigue Impact Scale (MFIS), a 21-item self-report questionnaire evaluating the impact of fatigue on physical, cognitive, and psychosocial functioning in individuals with multiple sclerosis. The total MFIS score ranges from 0 to 84, with higher scores indicating greater fatigue impact and worse fatigue-related outcomes. MFIS scores will be examined in relation to respiratory muscle strength and endurance.
Quality of Life (Multiple Sclerosis International Quality of Life Questionnaire) | Baseline
  Quality of life will be assessed using the Multiple Sclerosis International Quality of Life questionnaire (MusiQoL-31), a 31-item self-administered, multidimensional instrument specifically developed for individuals with multiple sclerosis. MusiQoL scores are linearly transformed to a 0-100 scale, with higher scores indicating better quality of life. MusiQoL-31 scores will be analyzed as clinical correlates of respiratory muscle strength and endurance.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail ÖZSOY, Assoc. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Zehra KORKUT, Assist. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Gülşah ÖZSOY, Assist. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Yasemin GEDİKLİ ERTÜRK, MSc. in PT, Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Selen GÜR ÖZMEN, Assoc. Prof. Dr., Study Chair — Bahçeşehir University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Istanbul, Türkiye; Haluk GÜMÜŞ, Prof. Dr., Study Chair — Selçuk University, Faculty of Medicine, Department of Neurology, Konya, Türkiye; Tuğbanur BAYTOK, Dr., Study Chair — Selçuk University, Faculty of Medicine, Department of Neurology, Konya, Türkiye; Cahit AYAN, Dr., Study Chair — Selçuk University, Faculty of Medicine, Department of Neurology, Konya, Türkiye
Locations (1):
- Selcuk University Faculty of Medicine Hospital MS Life Center, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bosnak-Guclu M, Gunduz AG, Nazliel B, Irkec C. Comparison of functional exercise capacity, pulmonary function and respiratory muscle strength in patients with multiple sclerosis with different disability levels and healthy controls. J Rehabil Med. 2012 Jan;44(1):80-6. doi: 10.2340/16501977-0900. PMID 22234321
- [Background] Mutluay FK, Gurses HN, Saip S. Effects of multiple sclerosis on respiratory functions. Clin Rehabil. 2005 Jun;19(4):426-32. doi: 10.1191/0269215505cr782oa. PMID 15929512
- [Background] Altintas A, Demir T, Ikitimur HD, Yildirim N. Pulmonary function in multiple sclerosis without any respiratory complaints. Clin Neurol Neurosurg. 2007 Apr;109(3):242-6. doi: 10.1016/j.clineuro.2006.09.004. Epub 2006 Oct 13. PMID 17046152
- [Background] Brown TR, Kraft GH. Exercise and rehabilitation for individuals with multiple sclerosis. Phys Med Rehabil Clin N Am. 2005 May;16(2):513-55. doi: 10.1016/j.pmr.2005.01.005. PMID 15893685
- [Background] Bishop M, Rumrill PD. Multiple sclerosis: Etiology, symptoms, incidence and prevalence, and implications for community living and employment. Work. 2015;52(4):725-34. doi: 10.3233/WOR-152200. PMID 26639011
- [Background] Tremlett H, Paty D, Devonshire V. Disability progression in multiple sclerosis is slower than previously reported. Neurology. 2006 Jan 24;66(2):172-7. doi: 10.1212/01.wnl.0000194259.90286.fe. PMID 16434648
- [Background] Calabresi PA. Diagnosis and management of multiple sclerosis. Am Fam Physician. 2004 Nov 15;70(10):1935-44. PMID 15571060
- [Background] Centonze D, Leocani L, Feys P. Advances in physical rehabilitation of multiple sclerosis. Curr Opin Neurol. 2020 Jun;33(3):255-261. doi: 10.1097/WCO.0000000000000816. PMID 32304436